CLINICAL TRIAL: NCT06515847
Title: A Study to Evaluate The Effects Of Nursing Care İmplementations Based On Kolcaba's Comfort Theory For The End Of Life Patients Comfort Levels and The Life Quality
Brief Title: Comfort and Quality of Life of Patients at the End of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Kadriye Nilay Genc, Assistant Professor , Dr Lecturer, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016.235.IRB2.117
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: End of Life
Keywords: Comfort; nurse; care
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kolcaba's nursing care plan (Experimental): While the patients of experimental group were cared according to the nursing care plan based on Kolcaba's comfort theory,
  Interventions: Other: End of Life Nursing Care Plan
- standard care plan (No Intervention): the patients of control group received the standard care plan of the institution

INTERVENTIONS:
Other: End of Life Nursing Care Plan — the patients of experimental group were cared according to the nursing care plan based on Kolcaba's comfort theory,
  Arms: Kolcaba's nursing care plan

SUMMARY:
A Research to Evaluate the Effect of Nursing Care Practices Based on Kolcaba's Comfort Theory on the Comfort Levels and Quality of Life of End-of-Life Patients.

Purpose: The study was carried out as a semi-experimental posttest with independent groups and a control group, in order to determine the effect of nursing care interventions on the patient's quality of life comfort level, based on Kolcaba's comfort theory. end-of-life patients.

Materials and Methods: This study compared 30 experimental and 30 control patients, aged between 25-70, at least primary school graduate, staying in the palliative care unit. He used the unit for at least two weeks and agreed to be part of this study. While the patients in the experimental group were cared for according to the nursing care plan based on Kolcaba's comfort theory, the patients in the control group were treated with the institution's standard care plan. The results were evaluated according to the standard comfort scale and the general quality of life scale.

ELIGIBILITY:
Inclusion Criteria:

* between 25-70 years old,
* communicable,
* at least primary school graduates,
* hospitalized in the unit for at least 2 weeks, and who agreed to participate in the study were included in the study.

Exclusion Criteria:

* All patients who did not meet the inclusion criteria and patients who were included in the study but died within 2 weeks were excluded from the study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Kolcaba's comfort theory | 2 week
  The general comfort scale scores of patients who are cared for according to the care plan prepared according to Kolcaba's comfort theory will be higher than the control group.
  The scale was developed by Kolcaba in 2006. Comfort includes the subscales of relief (9 items), relaxation (9 items) and overcoming problems (10 items). In evaluating the scale consisting of positive and negative items, negative items are reverse coded and summed. The average value is found by dividing the total score obtained by the number of scale items. The lowest possible value of 1 indicates low comfort, and the highest value of 6 indicates high comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahce University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study data will not be used for research by other researchers. It is specific to this study. Patient data will be kept confidential.